CLINICAL TRIAL: NCT01098175
Title: Peritoneal Cavity Conditioning During Open Surgery Decreases Postoperative Pain and Inflammation and Decreases Time to Restore Transit
Brief Title: Peritoneal Cavity Conditioning During Open Surgery.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Prof Philippe R. Koninckx, UZ Gasthuisberg, KULeuven
Other Study IDs: S52233
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Laparotomy; Thoracotomy
Keywords: laparotomy; thoracotomy; peritoneal conditioning; humidification; temperature control

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: open surgery with exposure of the surgical wound to the air.
- Full peritoneal conditioning: Full peritoneum cavity conditioning will be performed as follows. A continuous flow of less than 0.5 l/min of gas will be instilled in the lowest part of the operating wound. As gas premixed bottles with CO2+ 4% of oxygen and 10% of N2O will be used. This gas will be humidified and at 31-32 °C to be achieved by a commercial humidifier (Fisher and Paykel) programmed in order to maintain 100% relative humidity at 31-32°C upon entrance of the peritoneal cavity.

SUMMARY:
Given the observations in animal models and the available data in the human our hypothesis is that peritoneal cavity conditioning (carbon dioxide with 4% of oxygen and 10% of N2O, 100% humidification at 32°C,) during open surgery, will result in an important decrease in postoperative peritoneal inflammation, postoperative pain, and will restore bowel transit faster.

DETAILED DESCRIPTION:
Aim of the Trial :

RCT demonstrating that peritoneal cavity conditioning during open surgery will result in a less postoperative inflammation, less postoperative pain, and shorter time to flatus and transit.

ELIGIBILITY:
Inclusion criteria :

* patients will be stratified and randomised according to the type of surgery
* total laparoscopic hysterectomy,
* promontofixation
* cholecystectomy

Exclusion criteria :

* Any pre-existing condition increasing the risk of surgery such as age, pre-existing conditions as clotting disorders, heart or lung impairment etc.
* Not signed informed consent
* known allergic reaction to Sprayshield, Intercoat of hyalobarrier gel ® or - any bowel lesion requiring a single or double layer suture. (given that for none of the any anti-adhesion barriers safety has been proven following bowel lesions and suture)
* Any condition that might interfere with inflammatory parameters or pre-existing such as ,pregnancy, immunodeficiency, chronic inflammatory disease as Crohn's disease, chronic pain conditions as (peripheral neuropathy, pathology of the vertebral column and osteo-articular disease, any condition causing acute pain e.g. trauma.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Standard open surgery such as hysterectomy, cancer surgery, bowel resections, cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint : decreased pain on day 1 and 2 after surgery | 0 to 7 days
  Postoperative pain : will be assessed by visual analog scales (cfr Trial by Verguts & Koninckx, addendum I) assessed pain on day 1, 2 and 3 after surgery. Pain medication will be free, but preferentially ibuprofen will be used in order to permit easier comparison of pain killer intake.

SECONDARY OUTCOMES:
decrease in CRP and inflammatory parameters on day 1 and 2 or longer | day 1-4
  Postoperative inflammatory reaction : daily assessment of inflammatory parameters as CRP, leucocytosis , and temperature for 4 to 7 days are done routinely today.
  In some subsets of patients other more specific inflammatory parameters as Ca125, IL-6 can be investigated
lower peritoneal fluid volume on day 2 | day 2 after surgery
  Estimation of peritoneal fluid volume by ultrasound on the second day after surgery will be performed in some subsets of patients. We indeed recently validated a non-invasive and reliable assessment of peritoneal fluid volume by ultrasound. (Verguts et all, 2009) We expect that the postoperative peritoneal fluid volume will increase with the degree of peritoneal inflammation.
Shorter time to resumption of transit: time to first flatus and time to first stool | day1 to 5
  Time to first flatus and time to first stool will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: philippe R Koninckx, MD, Principal Investigator — UZ Gasthuisberg, KULeuven
Locations (1):
- UZ Gasthuisberg, Leuven, Belgium